CLINICAL TRIAL: NCT05560438
Title: Technology Assisted Rehabilitation for Upper Limb Function in Myotonic Dystrophy Type 1
Acronym: Technorehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Vikersund Rehabilitation Center (Unknown)
Responsible Party: Principal Investigator, Hilde Stendal Robinson, Professor, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 256361
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: Single subject experimental design (SSED) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technorehab (Experimental): Rehabilitation using Tyromotion Amadeo and Armeo Senso
  Interventions: Device: Tyromotion Amadeo and Armeo Senso

INTERVENTIONS:
Device: Tyromotion Amadeo and Armeo Senso — Robot assisted rehabilitation for arm- and hand function with Tyromotion Amadeo and Armeo Senso

SUMMARY:
Myotonic Dystrophy type 1 (DM1) is a genetic multisystem disease causing muscle weakness and myotonia. As a result, upper limb function might become impaired. There are little research regarding rehabilitation and exercise for upper limb function in DM1. It is known from research on lower limb function in DM1 and other muscular dystrophies, that there are possibilities to improve function also in these deteriorating diseases. In this single subject experimental design study, 6-10 adults with DM1, who are at an inpatient rehabilitation center, will get intensive, but personally adapted senso- and robot assisted rehabilitation for arm- and hand function with Tyromotion Amadeo and Armeo Senso. These devices have previously been used in rehabilitation research for other neurological conditions. The participants will be followed up, and evaluated at a weekly basis, using video consultations. Fine motor skill dexterity test (9HPT) and the Nut and Bolt test will be used, and active range of motion (ROM) and muscle strenght and movement of upper limb will be measured. Furthermore, patient reported outcome measures (PROMS) on hand impairment and myotonia will be used, all with purpose to evaluate upper limb function.

ELIGIBILITY:
Inclusion Criteria:

* Granted rehabilitation at Vikersund Rehabilitation center Genetical confirmed myotonic dystrophy diagnosis MIRS score between 2-5

Exclusion Criteria:

* MIRS score on 1 Reduced Cognitive function and unable to participate in technological rehabilitation and digital evaluation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fine motor skill dexterity test, 9 hole peg test (9HPT) | 1-3 minutes
  Motor skill test

SECONDARY OUTCOMES:
Range of motion (ROM) | 5-10 minutes
  Measure of ROM in upper limb joints
Nut and Bolt test | 5 minutes
  Motor skill test
Hand strength | 5 minutes
  Measured by Jamar digital dynamometer
Pinch Gauge | 5 minutes
  Finger strength measures by Jamar digital pinch gauge

OTHER OUTCOMES:
Abilhand | 5 minutes
  Patient reported outcome measure, measure of manual ability for adults with upper limb impairment
Myotonia behavior scale | 1-5 minutes
  Patient reported outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Stendal Robinson, PhD, Principal Investigator — University of Oslo
Locations (1):
- Vikersund Rehabilitation Center, Vikersund, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
This is a single subject experimental design study, and the data will not be available for other researchers. This is to protect the participants identity.